CLINICAL TRIAL: NCT01430585
Title: An Open-Label, Randomised Phase 1b/2 Study Of PF-04691502 In Combination With Letrozole Compared With Letrozole Alone In Patients With Estrogen Receptor Positive, Her-2 Negative Early Breast Cancer
Brief Title: Pre-Operative Study of PF-4691502 With Letrozole Compared To Letrozole Alone In Patients With Early Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1271003
Record Dates: First submitted 2011-08-18; First posted 2011-09-08 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-07

CONDITIONS: Early Breast Cancer (Phase 2); Advanced Breast Cancer (Phase 1b)
Keywords: Ki-67; postmenopausal early breast cancer; ER positive/HER2 negative early breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 2-amino-8-(4-(2-hydroxyethoxy)cyclohexyl)-6-(6-methoxypyridin-3-yl)-4-methylpyrido(2,3-d)pyrimidin-7(8H)-one; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: PF-04691502
- B (Experimental)
  Interventions: Drug: PF-04691502 in combination with Letrozole
- C (Active Comparator)
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: PF-04691502 — PF-04691502 administered as single agent for 2 weeks. After this period, patients in this arm will take PF-04691502 in combination with Letrozole until Week 6. Beyond Week 6, if considered appropriate, patients can be treated with the combination for up to 10 additional weeks until breast surgery.
  Arms: A
Drug: PF-04691502 in combination with Letrozole — PF-04691502 in combination with Letrozole will be administered for 6 weeks. Beyond Week 6, if considered appropriate, patients can be treated for up to 10 additional weeks until breast surgery.
  Arms: B
Drug: Letrozole — Letrozole will be administered for 6 weeks. Beyond Week 6, if considered appropriate, patients can be treated for up to 10 additional weeks until breast surgery.
  Arms: C

SUMMARY:
PF-04691502 is an inhibitor of PI3K and mTOR kinase. Published data support the hypothesis that a PI3K/mTOR antagonist in combination with letrozole might mitigate the intrinsic or acquired resistance to hormonal therapy and restore hormone sensitivity in high risk (high Ki-67) patient population of hormone-sensitive breast cancers. In addition, Ki-67, a marker of cellular proliferation, could be used to select those patients who benefit from treatment with a PI3K-pathway inhibitor.

DETAILED DESCRIPTION:
The study was prematurely discontinued on 09Oct2012 due to the tolerability findings in 2 clinical studies testing PF-04691502 that have prompted the Sponsor to re-evaluate the strategic goals of the program. In the study B1271003 an unexpected frequency of severe skin toxicity was observed and in the study B1271004 5 cases of drug induced pneumonitis were reported.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1 - Postmenopausal women with diagnosis of breast cancer, metastatic disease or locally advanced disease / Estrogen Receptor positive and HER-2 negative / candidate to receive Letrozole
* Phase 2 - Postmenopausal women with newly diagnosed primary breast cancer / Estrogen Receptor positive and HER-2 negative / Ki-67 levels >10% positive cells
* Phase 1 & 2 - Glucose control, adequate bone marrow, liver, renal, and cardiac function

Exclusion Criteria:

* Inflammatory carcinoma / Prior therapy with an agent active on PI3K and/or mTOR / Significant gastrointestinal abnormalities, which may impair intake, transit or absorption of the study drugs / Current or anticipated need for food or drugs that are known inhibitors or inducers of CYP3A4

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Pfizer Investigational Site, Charleroi, Belgium
- Pfizer Investigational Site, Milan, Italy
- Pfizer Investigational Site, Barcelona, Barcelona, Spain
- Sweden (2):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Stockholm

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1271003&StudyName=Pre-Operative%20Study%20of%20PF-4691502%20With%20Letrozole%20Compared%20To%20Letrozole%20Alone%20In%20Patients%20With%20Early%20Breast%20Cancer%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to premature termination of the study, the planned treatments of Phase 2, PF-04691502, then PF-04691502 + Letrozole (Phase 2), PF-04691502 + Letrozole (Phase 2) and Letrozole (Phase 2), were not administered.
Groups:
- PF-04691502 + Letrozole (Phase 1B): Letrozole 2.5 milligram (mg) tablet orally on Day 1 followed by PF-04691502 8 mg tablet orally once daily from Day 2 until Day 11 and then a combination of PF-04691502 8 mg tablet and letrozole 2.5 mg tablet orally once daily from Day 12 until progression of disease, occurrence of unacceptable toxicity or withdrawal of consent. Dose of PF-04691502 was reduced to 6 mg orally once daily based on preliminary safety analysis conducted in the first 7 participants evaluable for safety.
Period: Overall Study
Arm/Group | PF-04691502 + Letrozole (Phase 1B)
Started | 14
Completed | 0
Not Completed | 14
Not completed — Death | 1
Not completed — Objective Progression or Relapse | 3
Not completed — Study Terminated by Sponsor | 3
Not completed — Other | 7

BASELINE CHARACTERISTICS:
Arm/Group | PF-04691502 + Letrozole (Phase 1B)
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 60.5 [51 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs): Phase 1B
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. SAE: an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study treatment and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Phase 1B: Baseline up to 28 days after last administration of study treatment
Population: Safety analysis set included all enrolled participants who started study treatment.
Measure: Number; unit: participants
Arm/Group | PF-04691502 + Letrozole (Phase 1B)
Number analyzed (Participants) | 14
participants
  SAEs | 7
  AEs | 14

2. Primary Outcome: Change From Baseline in Ki-67 Percent Positive Tumor Cells in Biopsied Tumor Tissue at Week 6: Phase 2
Description: Nuclear proliferation marker Ki-67 was to be assessed by immunohistochemistry technique in all specimens.
Time Frame: Phase 2: Baseline, Week 6
Population: Data was not analyzed due to premature termination of the study. No participant was enrolled in phase 2 of the study.
Groups:
- PF-04691502, Then PF-04691502 + Letrozole (Phase 2): PF-04691502 6 mg tablet orally once daily up to Week 2 followed by combination of PF-04691502 6 mg tablet and letrozole 2.5 mg tablet orally once daily up to Week 6 or 16 as per investigator's discretion.
- PF-04691502 + Letrozole (Phase 2): Combination of PF-04691502 6 mg tablet and letrozole 2.5 mg tablet orally once daily up to Week 6 or 16 as per investigator's discretion.
- Letrozole (Phase 2): Letrozole 2.5 mg tablet orally once daily up to Week 6 or 16 as per investigator's discretion.
Arm/Group | PF-04691502, Then PF-04691502 + Letrozole (Phase 2) | PF-04691502 + Letrozole (Phase 2) | Letrozole (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs): Phase 2
Description: as for outcome 1
Time Frame: Phase 2: Baseline up to 28 days after last administration of study treatment
Population: Data was not analyzed due to premature termination of the study. No participant was enrolled in phase 2 of the study.
Arm/Group | PF-04691502, Then PF-04691502 + Letrozole (Phase 2) | PF-04691502 + Letrozole (Phase 2) | Letrozole (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Tests Abnormalities: Phase 1B and 2
Description: Laboratory analysis planned to include blood chemistry, hematology and urinalysis.
Time Frame: Phase 1B: Baseline up to end of treatment (Week 34); Phase 2: Baseline up to Week 16 or early termination (ET)
Population: Data was not analyzed due to premature termination of the study. No participant was enrolled in phase 2 of the study.
Arm/Group | PF-04691502 + Letrozole (Phase 1B) | PF-04691502, Then PF-04691502 + Letrozole (Phase 2) | PF-04691502 + Letrozole (Phase 2) | Letrozole (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs: Phase 1B and 2
Description: Vital signs assessments planned to include measurement of blood pressure and heart rate.
Time Frame: Phase 1B: Baseline up to 28 days after last dose of study treatment (Week 34); Phase 2: Baseline up to Week 16 or ET
Population: Data was not analyzed due to premature termination of the study. No participant was enrolled in phase 2 of the study.
Arm/Group | PF-04691502 + Letrozole (Phase 1B) | PF-04691502, Then PF-04691502 + Letrozole (Phase 2) | PF-04691502 + Letrozole (Phase 2) | Letrozole (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Corrected QT (QTc) Interval: Phase 1B
Time Frame: Phase 1B: Baseline up to end of treatment (Week 34)
Population: Data was not analyzed due to premature termination of the study.
Arm/Group | PF-04691502 + Letrozole (Phase 1B)
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With Objective Response (OR): Phase 1B and 2
Description: Number of participants with objective response based on assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR was defined as complete disappearance of all target lesions and non-target lesions, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis less than [<] 10 millimeter [mm]). No appearance of new lesions and normalization of tumor marker levels. PR was defined as greater than or equal to (>=) 30 percent (%) decrease from baseline of the sum of diameters of all target lesions, using the short diameter in the sum for target nodes and the longest diameter in the sum for all other target lesions.
Time Frame: Phase 1B: Baseline, Week 12, end of treatment (Week 34); Phase 2: Baseline, Week 6, 16 or ET
Population: Data for phase 1B was reported in individual participant listings but not statistically summarized for analysis due to premature termination of the study. No participant was enrolled in phase 2 of the study.
Arm/Group | PF-04691502 + Letrozole (Phase 1B) | PF-04691502, Then PF-04691502 + Letrozole (Phase 2) | PF-04691502 + Letrozole (Phase 2) | Letrozole (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Pharmacokinetic (PK) Parameters of PF-04691502 and Letrozole: Phase 1B and 2
Description: Phase 1B: Following PK parameters were planned to be calculated from the plasma concentration time data using standard non-compartmental methods. For PF-04691502: area under the curve from time zero to last quantifiable concentration (AUClast), area under the curve from time zero to end of dosing interval (AUCtau), maximum observed plasma concentration (Cmax), minimum observed plasma trough concentration (Cmin), average plasma concentration (Cavg), time to reach maximum observed plasma concentration (Tmax), observed accumulation ratio (Rac [obs]); for letrozole: AUClast, Cmax. Phase 2: Following PK parameters were planned to be calculated for PF-04691502 from the plasma concentration time data using standard non-compartmental methods- AUClast, Cmax and Tmax.
Time Frame: Phase 1B: 0 (pre-dose), 1, 2, 4, 6, 24 hours on Day 1 (letrozole alone), Day 2 (PF-0491502 alone), Day 12, Week 5 (PF-0491502 and letrozole in combination); Phase 2: 0 (pre-dose), 1, 2, 4, 6, 24 hours on Day 1, pre-dose on Week 2, 6
Population: as for outcome 7
Arm/Group | PF-04691502 + Letrozole (Phase 1B) | PF-04691502, Then PF-04691502 + Letrozole (Phase 2) | PF-04691502 + Letrozole (Phase 2) | Letrozole (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline in Pharmacodynamic, Cell Proliferation and Survival Biomarkers in Biopsied Tumor Tissue at Week 2 and 6: Phase 2
Description: Change from baseline in following pharmacodynamic parameters were planned to be calculated: expression and/or phosphorylation of Phosphoinositide-3-kinase (PI3K) pathway proteins in biopsied tumor tissue and markers of cell cycle and survival.
Time Frame: Phase 2: Baseline, Week 2, 6
Population: Data was not analyzed due to premature termination of the study. No participant was enrolled in phase 2 of the study.
Arm/Group | PF-04691502, Then PF-04691502 + Letrozole (Phase 2) | PF-04691502 + Letrozole (Phase 2) | Letrozole (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Genetic Alterations: Phase 2
Description: Following genetic alterations were planned to be analyzed: mutations in Phosphoinositide 3-kinase, catalytic, alpha (PIK3CA), amplification of PIK3CA, Phosphate and tensin homolog (PTEN) deficiency, and changes in other genes or proteins in, or impacting V-Ki-ras2 Kirsten Rat Sarcoma Viral Oncogene Homolog (KRAS), Insulin-like Growth Factor 1 Receptor (IGF-1R), phosphatidylinositol 3-kinase (PI3K)/ mammalian target of rapamycin (mTOR) pathway.
Time Frame: Phase 2: Baseline, Week 2, 6
Population: Data was not analyzed due to premature termination of the study. No participant was enrolled in phase 2 of the study.
Arm/Group | PF-04691502, Then PF-04691502 + Letrozole (Phase 2) | PF-04691502 + Letrozole (Phase 2) | Letrozole (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-04691502 + Letrozole (Phase 1B)
Serious Adverse Events (participants affected / at risk) | 7/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04691502 + Letrozole (Phase 1B) (N=14)
Rash (Skin and subcutaneous tissue disorders) | 2
Rash maculo (Skin and subcutaneous tissue disorders) | 2
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Disease progression (General disorders) | 1
General physical health deterioration (General disorders) | 1
Pyrexia (General disorders) | 1
Lung infection (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04691502 + Letrozole (Phase 1B) (N=14)
Diarrhoea (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 7
Stomatitis (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Oral discomfort (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 6
Asthenia (General disorders) | 3
Chills (General disorders) | 3
Mucosal inflammation (General disorders) | 3
Catheter site related reaction (General disorders) | 1
Early satiety (General disorders) | 1
General physical health deterioration (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 8
Decreased appetite (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Fluid retention (Metabolism and nutrition disorders) | 1
Folate deficiency (Metabolism and nutrition disorders) | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Urinary tract infection (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 2
Asymptomatic bacteriuria (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Oral fungal infection (Infections and infestations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Blood creatinine increased (Investigations) | 2
Blood insulin increased (Investigations) | 2
Weight decreased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood urine present (Investigations) | 1
Platelet count decreased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Hot flush (Vascular disorders) | 2
Lymphoedema (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Varicose vein (Vascular disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Polycythaemia (Blood and lymphatic system disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Oliguria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Agitation (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Conjunctivitis (Eye disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1

LIMITATIONS AND CAVEATS:
Study was prematurely terminated due to PF-04691502 tolerability findings that prompted Sponsor to re-evaluate strategic goals of program. Unexpected frequency of severe skin toxicity was observed and no participant was enrolled in phase 2 of study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.